CLINICAL TRIAL: NCT01397955
Title: Drug Use Investigation of Julina Tablets 0.5 mg (Postmenopausal Osteoporosis)
Brief Title: Julina Post-marketing Surveillance for Postmenopausal Osteoporosis in Japan
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15075
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: Julina; Postmenopausal osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Drug (incl. Placebo)
  Interventions: Drug: E2 transdermal (Julina, BAY86-5435)

INTERVENTIONS:
Drug: E2 transdermal (Julina, BAY86-5435) — Patients in daily life treatment receiving Julina for postmenopausal osteoporosis

SUMMARY:
This study is a regulatory post-marketing surveillance in Japan, and it is a local prospective and observational study of patients who have received Julina for postmenopausal osteoporosis. The objective of this study is to assess safety and efficacy of using Julina in clinical practice. A total 100 patients will be recruited and followed 3 years since starting Julina administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received Julina for postmenopausal osteoporosis

Exclusion Criteria:

* Patients who are contraindicated based on the product label

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population of this study is patients who have received a prescription of Julina on the basis of the decision of the treating gynecologist. The study is expected to collect data of 100 patients in about 20 gynecological practices in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2009-01; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions and serious adverse events in subject who received Julina | After Julina administration, upto 3 years

SECONDARY OUTCOMES:
Incidence of adverse drug reactions in subpopulation with baseline data (such as demographic data, concomitant disease, hysterectomy) and dose of Julina | At baseline and after Julina administration, upto 3 years
Effectiveness evaluation assessment by the three rank scales: improvement, not changed, and worse | At baseline and at end of Julina treatment, upto 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Japan